CLINICAL TRIAL: NCT04974814
Title: Comparison of the Treatment Efficacy of Rosuvastatin Versus Atorvastatin Loading Prior to Percutaneous Coronary Intervention in ST-Segment Elevation Myocardial Infarction
Brief Title: Effect of Statin Preloading in STEMI in Improving PCI Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Esraa M. Adel, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: statin in STEMI
Record Dates: First submitted 2021-07-06; First posted 2021-07-23 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: STEMI; statin; PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Intervention Model Description: The clinical study will be a prospective open label randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): in this group patients will not receive statin before primary PCI
  Interventions: Drug: Control Test
- atorvastatin group (Active Comparator): in this group patients will receive 80 mg atorvastatin single dose before primary PCI
  Interventions: Drug: Atorvastatin 80mg
- rosuvastatin group (Active Comparator): in this group patients will receive 40 mg rosuvastatin single dose before primary PCI
  Interventions: Drug: Rosuvastatin 40mg

INTERVENTIONS:
Drug: Rosuvastatin 40mg — patients in active arms will be preloaded with a single 40 mg rosuvastatin in ER before PCI
  Arms: rosuvastatin group
Drug: Atorvastatin 80mg — patients in active arms will be preloaded with a single 80 mg atorvastatin in ER before PCI
  Arms: atorvastatin group
Drug: Control Test — patients in control arm will not preloaded with statin in ER before PCI
  Arms: control group

SUMMARY:
To compare the effect of a single high dose of atorvastatin versus rosuvastatin preloading on microvascular coronary perfusion as determined by CTFC in patients with ST-segment elevation myocardial infarction (STEMI) undergoing PCI.

DETAILED DESCRIPTION:
Acute myocardial infarction (MI) indicates irreversible myocardial injury resulting in necrosis of a significant portion of myocardium which is caused mostly by coronary plaque rupture or erosion. It could result in several clinical complications and impact cardiac prognosis .

Worldwide, ischemic heart disease is the single most common cause of death and its frequency is increasing, now Accounts for almost 1.8 million annual deaths.

Cholesterol reduction with HMG-CoA (3-hydroxy-3-methylglutaryl coenzyme A) reductase inhibitors or statins has been shown to improve mortality and cardiovascular morbidity in patients with established coronary artery disease (CAD).

Previous evidence suggests that statins have various favorable effects on vascular system that are not directly related to their impact on lipid metabolism. Beyond lowering lipids, statins have favorable effects on platelet adhesion, thrombosis, endothelial function, plaque stability, and inflammation. . As with ACS, the vascular injury from coronary angioplasty and stent placement induces platelet activation, thrombosis, and inflammation within the vessel wall and the distal microvasculature. Therefore, in addition to a long-term benefit associated with lipid lowering, statin therapy might play a beneficial role early after PCI.

Conventional TIMI flow grading (Thrombolysis In Myocardial Infarction) is a predictor of cardiac outcome after acute myocardial infarction and PCI, but it has several limitations.

The CTFC (corrected TIMI frame count) another approach to grade flow impairment, is an objective, quantitative, reproducible, and sensitive index for coronary blood flow[9].

TIMI flow may appear normal visually, but may correlate to abnormal CTFC. The CTFC has been proposed to have incremental prognostic accuracy in predicting survival outcome with reperfusion therapy . Higher CTFC values after PCI have also been found to be associated with poor clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The Presence of symptoms (<12h).
* ST-segment elevation of at least 0.1Mv in two contiguous leads of electrocardiogram or new onset left bundle branch block.
* Patients age 18 to 80 years.

Exclusion Criteria:

* Previous (within 3 months) or current treatment with statins.
* Known allergy to heparin, aspirin, clopidogrel, or abciximab.
* Active severe bleeding.
* Pregnancy.
* History of major surgery or trauma.
* Significant gastrointestinal or genitourinary bleeding (<6 weeks).
* History of cerebrovascular attack (within 2 years) or cerebrovascular attack with a significant residual neurological deficit.
* Cardiogenic shock with mechanical ventilation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
angiographic parameters | 3 months
  CTFC (corrected TIMI frame count) In the CTFC method, the number of frames required for dye to reach a standardized distal landmark is counted. A correction factor is required to compensate for the longer length of the left anterior descending artery (LAD) compared with the circumflex and right coronary arteries (the number of frames required for dye to traverse the LAD is divided by 1.7). The frame count number after adjustment for vessel length is given the term 'corrected TIMI frame count'.
STR (ST-segment resolution) (STR) | 3 months
  ST-segment resolution (STR) was calculated as the sum of ST-segment elevation on initial ECG minus the sum of ST-segment elevation on the ECG at 90 min after PCI, divided by the sum of ST- segment elevation on initial ECG, and was expressed as a percentage . The complete early STR was defined as more than or equal to 70% STR.

CONTACTS AND LOCATIONS:
Overall Officials: Esraa M Adel, bachelor, Principal Investigator — National Heart Institute; Ahmed A El berry, phd, Study Director — Beni-Suef University; Raghda R Hussein, phd, Study Director — Beni-Suef University; Ahmed A Abd el hamid, Study Director — National Heart Institute
Locations (1):
- National Heart Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elserafy AS, Farag NM, El Desoky AI, Eletriby KA. Effect of high-intensity statin preloading on TIMI flow in patients presenting with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention. Egypt Heart J. 2020 Jul 10;72(1):40. doi: 10.1186/s43044-020-00074-0. PMID 32651772
- [Result] Jang Y, Zhu J, Ge J, Kim YJ, Ji C, Lam W. Preloading with atorvastatin before percutaneous coronary intervention in statin-naive Asian patients with non-ST elevation acute coronary syndromes: A randomized study. J Cardiol. 2014 May;63(5):335-43. doi: 10.1016/j.jjcc.2013.09.012. Epub 2013 Nov 9. PMID 24216317
- [Result] Ma M, Bu L, Shi L, Guo R, Yang B, Cao H, Luo L, Lu L. Effect of loading dose of atorvastatin therapy prior to percutaneous coronary intervention in patients with acute coronary syndrome: a meta-analysis of six randomized controlled trials. Drug Des Devel Ther. 2019 Apr 16;13:1233-1240. doi: 10.2147/DDDT.S196588. eCollection 2019. PMID 31354240